CLINICAL TRIAL: NCT02574598
Title: A Randomized Crossover, Phase II Clinical Trial of MK-3475 in Combination With Docetaxel Versus Docetaxel Alone in Patients With Non-Small Cell Lung Cancer (NSCLC) Previously Treated.
Brief Title: MK-3475 in Combination With Docetaxel vs Docetaxel Alone in Non-Small Cell Lung Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Instituto Nacional de Cancerologia de Mexico (Other)
Responsible Party: Principal Investigator, Oscar Gerardo Arrieta Rodríguez, Investigador en Ciencias Médicas "E", Instituto Nacional de Cancerologia de Mexico
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INCAN/014/033/ICI; INCAN/014/033/ICI (Other: National Cancer Institute of Mexico)
Record Dates: First submitted 2015-10-09; First posted 2015-10-14 (Estimated); Results first posted 2020-12-14 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2020-12

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: PDL1; monoclonal antibody
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab; Docetaxel

STUDY DESIGN:
Intervention Model Description: Patients will be randomly assigned (1:1) using a random numbers table to receive either monotherapy Docetaxel for 6 cycles or Pembrolizuymab plus Docetaxel for 6 cycles, following with maintenance therapy with Pembrolizumab until disease progression or unacceptable toxicity.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Docetaxel + MK-3475 (Experimental): Docetaxel 75 mg/m2 every 3 weeks until progression of disease
  MK-3475 (administered on day 8) 200mg every 3 until progression of disease
  Interventions: Drug: MK-3475; Drug: Docetaxel
- Docetaxel (Active Comparator): Docetaxel 75 mg/m2 every 3 weeks until progression of disease followed by MK-3475 200mg every 3 until progression of disease
  Interventions: Drug: MK-3475; Drug: Docetaxel

INTERVENTIONS:
Drug: MK-3475 — The dosing interval of pembrolizumab can be increased in case of toxicity.
  Other Names: pembrolizumab
Drug: Docetaxel — Use on both arms as standard of care.
  Other Names: taxotere

SUMMARY:
This is a phase II open-label randomized clinical trial of MK-3475 (Pembrolizumab) on previously treated non-small cell lung cancer (NSCLC) patients . This drug has shown to allow partial response according to the immune-related response criteria and the response evaluation criteria in solid tumors (RECIST). The main endpoint is to compare the overall response rate (ORR) of MK-3475 with docetaxel or docetaxel alone in patients with advanced NSCLC.

DETAILED DESCRIPTION:
MK-3475 (MK-3475) is an IgG4 monoclonal antibody to PD1, which received a 'breakthrough therapy' designation for advanced melanoma from the FDA in January 2013. Preliminary results from the NSCLC cohort of a phase I dose expansion trial of MK-3475 were presented at the 2013 World Conference on Lung Cancer meeting. MK-3475 was administered intravenously every three weeks, and continued until disease progression based upon immune related response criteria (irRC) or unacceptable toxicity. IrRC take into account the potential for different patterns of response that can be seen with immunotherapy. Of the 38 patients with previously treated advanced NSCLC evaluable for efficacy, 9 (24 percent) achieved at least partial response by irRC. Standard oncology criteria for response (Response Evaluation Criteria In Solid Tumors, RECIST were available for 33 of these patients, with at least a partial response in seven patients (21 percent). Median overall survival was 51 weeks. Therapy was well tolerated, with one case of pneumonitis (grade 2) and one case of pulmonary edema (grade 3) reported. Tumor PDL1 expression (assessed with a different assay than that used for the trials evaluating Nivolumab and MPDL3280A; antibody used undisclosed) was available for 33 of the patients who had irRC assessments and 29 of those with standard oncology (RECIST) assessment. Of the 9 patients with PDL1 positivity and irRC response data, 6 achieved at least partial response (67 percent); of the 7 patients with PDL1 positivity and standard oncology response data, 4 achieved response (57 percent). Of note, 1 of 24 patients with PDL1 negativity achieved response by irRC; 2 of 22 patients with PDL1 negativity had response by standard oncology criteria (RECIST).

Based upon these results, a randomized phase II trial comparing MK-3475 to standard salvage docetaxel in patients with advanced NSCLC has been launched (NCT01905657), however there is no study in which the synergistic activity of Docetaxel + MK-3475 were evaluated, this could open the possibility of using this drug concurrently with Docetaxel as standard therapy in patients with progression of the disease despite a double platinum-based regimen.

Measure the expression levels of PD1/PD-L1/PD-L2 subpopulations tumor cells of patients with NSCLC who come to the clinic of the National Cancer Institute and relevant way, associating their role forecast and its potential as a biomarker, relating the PD-L1 levels with clinicopathologic characteristics of the patients studied.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent

   1. Patients should be signed and dated form of written informed consent approved by the IRB / IEC in accordance with regulatory and institutional guidelines. This must be obtained before performing any procedure related to the protocol that are not part of the normal care of the patient.
   2. Patients must be willing and able to comply with scheduled visits , treatment program , laboratory testing including filling of questionnaires the results reported by the patient and other study requirements .
2. Target Population

   1. Subjects with locally advanced NSCLC of squamous cell and non-squamous cell (adenocarcinoma and big cells) histological or cytologically documented , those who submit Stage IIIB / IV or recurrent disease after receiving radiation treatment or surgical resection
   2. Men and women ≥ 18 years of age.
   3. Performance status Eastern Cooperative Oncology Group ( ECOG ) ≤ 1.
   4. Subjects must have measurable disease by CT or MRI according to RECIST 1.1 criteria Radiographic Evaluation of Tumor on in the span of 28 days before randomization.
   5. The target lesions may be located on a previously irradiated field exists if documented progression of disease (radiographic) in that site. Subjects progression or recurrence of the disease must have experienced during or after prior chemotherapy regimen containing platinum in metastatic disease.

      This includes individuals who meet the following criteria:
      1. Subjects who received pemetrexed, bevacizumab or erlotinib as maintenance therapy (non-progressors double platinum-based chemotherapy) and progressed are eligible However, patients who received a wild EGFR tyrosine kinase inhibitor after failure of prior platinum-based therapy were excluded.
      2. Eligible patients who received double- platinum -based chemotherapy in adjuvant or neo adjuvant (after surgery and / or radiation) and developed recurrent or metastatic disease within 6 months after treatment ends
      3. Eligible individuals with recurrent disease > 6 months after adjuvant chemotherapy or neoadjuvant platinum-based , who also subsequently progressed during or after one platinum-based doublet regimen to treat recurrences
      4. Subjects with a known mutation of EGFR and received EGFR TKI (erlotinib , gefitinib or experimental) and double platinum-based chemotherapy ( regardless of the order of administration).
      5. subjects with known ALK translocation double receiving platinum-based chemotherapy and ALK inhibitor ( crizotinib or experimental )
      6. patients who have received >30Gy to the chest should have waited at least 6 months from completing radiation to starting pembrolizumab.
   6. must be available a blood sample, for evaluation of biomarkers. Samples must be received by the central laboratory before randomization.
   7. All baseline laboratory requirements will be evaluated , and must be obtained -14 days of randomization. The screening laboratory values must meet the following criteria:

   i) WBC ≥ 2000/μL ii) iNeutrophils ≥ 1500/μL iii) Platelets ≥ 100 x 10 ³ / uL iv) Hemoglobin ≥ 9.0 g / dL v) Serum creatinine ≤ 1.5 x ULN or creatinine clearance > 40 mL / min (using the Cockcroft / Gault ) Women : CrCl = (140 - age in years) x weight in kg x 0.85 72 x serum creatinine in mg / dL Males: CrCl = (140 - age in years) x weight in kg x 1.00 72 x serum creatinine in mg / dL vi) ≤ 1.5 X ULN AST vii) ≤ 1.5 X ULN ALT viii) Total bilirubin ≤ 1.5x ULN (except for subjects with Gilbert 's Syndrome who must have total bilirubin < 3.0 mg / dL ) h ) pretreatment with radiotherapy or radiosurgery at least 3 weeks must be completed before randomization.

   i ) Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
3. Age and Reproductive Status

   1. Women with reproductive potential ( WOCBP ) should use contraceptive methods based on tables found in Appendix 2 . When a teratogenic drug test is used , and / or a drug for which there is not enough information to assess teratogenicity ( have not been conducted preclinical studies) are required to use a highly effective method of contraception ( failure rate less than 1 % per year). Individual methods of contraception should be determined in consultation with the researcher.
   2. The WOCBP must have a negative pregnancy test in serum or urine ( minimum sensitivity 25 IU / L or equivalent units of HCG ) 24 hours before starting the investigational product .
   3. Women should not be breastfeeding .
4. Subjects must:

   1. Be willing and able to provide written informed consent/assent for the trial.
   2. Be > 18 years of age on day of signing informed consent.
   3. Have measurable disease based on RECIST 1.1.
   4. Have provided tissue from an archival tissue sample or newly obtained core or excisional biopsy of a tumor lesion.
   5. Have a performance status of 0 or 1 on the ECOG Performance Scale.

6. Demonstrate adequate organ function as defined in Table 1, all screening labs should be performed within 10 days of treatment initiation.

Exclusion Criteria:

The subject must be excluded from participating in the trial if the subject:

1. Is currently participating in or has participated in a study of an investigational agent or using an investigational device within 4 weeks of the first dose of treatment.
2. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
3. Has had a prior monoclonal antibody within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
4. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.

   * Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.
   * Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
5. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy.
6. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment.
7. Has an active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents. Subjects with vitiligo or resolved childhood asthma/atopy would be an exception to this rule. Subjects that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study. Subjects with hypothyroidism stable on hormone replacement or Sjorgen's syndrome will not be excluded from the study.
8. Has evidence of interstitial lung disease or active, non-infectious pneumonitis.
9. Has an active infection requiring systemic therapy.
10. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
11. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
12. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
13. Has received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-Cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways).
14. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
15. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
16. Has received a live vaccine within 30 days prior to the first dose of trial treatment.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2016-06; Primary Completion 2019-10 (Actual); Study Completion 2020-11-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Oscar G Arrieta, MD, MSc, Principal Investigator — National Institute of Cancer of Mexico
Locations (1):
- National Cancer Institute of Mexico, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD, all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Once the information recruitment is concluded ( starting 6 months after publication)
Access Criteria: Only information will be given to the principal investigator, with a signed request and registration of the protocol.
  For research and statistical purposes that are required. For future statistics publications related to this study.

REFERENCES:
- [Background] Disis ML. Immune regulation of cancer. J Clin Oncol. 2010 Oct 10;28(29):4531-8. doi: 10.1200/JCO.2009.27.2146. Epub 2010 Jun 1. PMID 20516428
- [Background] Dong H, Strome SE, Salomao DR, Tamura H, Hirano F, Flies DB, Roche PC, Lu J, Zhu G, Tamada K, Lennon VA, Celis E, Chen L. Tumor-associated B7-H1 promotes T-cell apoptosis: a potential mechanism of immune evasion. Nat Med. 2002 Aug;8(8):793-800. doi: 10.1038/nm730. Epub 2002 Jun 24. PMID 12091876
- [Background] Sharpe AH, Freeman GJ. The B7-CD28 superfamily. Nat Rev Immunol. 2002 Feb;2(2):116-26. doi: 10.1038/nri727. PMID 11910893
- [Background] Brown JA, Dorfman DM, Ma FR, Sullivan EL, Munoz O, Wood CR, Greenfield EA, Freeman GJ. Blockade of programmed death-1 ligands on dendritic cells enhances T cell activation and cytokine production. J Immunol. 2003 Feb 1;170(3):1257-66. doi: 10.4049/jimmunol.170.3.1257. PMID 12538684
- [Background] Francisco LM, Sage PT, Sharpe AH. The PD-1 pathway in tolerance and autoimmunity. Immunol Rev. 2010 Jul;236:219-42. doi: 10.1111/j.1600-065X.2010.00923.x. PMID 20636820
- [Background] Deschoolmeester V, Baay M, Van Marck E, Weyler J, Vermeulen P, Lardon F, Vermorken JB. Tumor infiltrating lymphocytes: an intriguing player in the survival of colorectal cancer patients. BMC Immunol. 2010 Apr 12;11:19. doi: 10.1186/1471-2172-11-19. PMID 20385003
- [Background] Liotta F, Gacci M, Frosali F, Querci V, Vittori G, Lapini A, Santarlasci V, Serni S, Cosmi L, Maggi L, Angeli R, Mazzinghi B, Romagnani P, Maggi E, Carini M, Romagnani S, Annunziato F. Frequency of regulatory T cells in peripheral blood and in tumour-infiltrating lymphocytes correlates with poor prognosis in renal cell carcinoma. BJU Int. 2011 May;107(9):1500-6. doi: 10.1111/j.1464-410X.2010.09555.x. Epub 2010 Aug 24. PMID 20735382
- [Background] Polcher M, Braun M, Friedrichs N, Rudlowski C, Bercht E, Fimmers R, Sauerwald A, Keyver-Paik MD, Kubler K, Buttner R, Kuhn WC, Hernando JJ. Foxp3(+) cell infiltration and granzyme B(+)/Foxp3(+) cell ratio are associated with outcome in neoadjuvant chemotherapy-treated ovarian carcinoma. Cancer Immunol Immunother. 2010 Jun;59(6):909-19. doi: 10.1007/s00262-010-0817-1. Epub 2010 Jan 20. PMID 20087581
- [Background] Topalian SL, Hodi FS, Brahmer JR, Gettinger SN, Smith DC, McDermott DF, Powderly JD, Carvajal RD, Sosman JA, Atkins MB, Leming PD, Spigel DR, Antonia SJ, Horn L, Drake CG, Pardoll DM, Chen L, Sharfman WH, Anders RA, Taube JM, McMiller TL, Xu H, Korman AJ, Jure-Kunkel M, Agrawal S, McDonald D, Kollia GD, Gupta A, Wigginton JM, Sznol M. Safety, activity, and immune correlates of anti-PD-1 antibody in cancer. N Engl J Med. 2012 Jun 28;366(26):2443-54. doi: 10.1056/NEJMoa1200690. Epub 2012 Jun 2. PMID 22658127
- [Background] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774
- [Background] Wolchok JD, Hoos A, O'Day S, Weber JS, Hamid O, Lebbe C, Maio M, Binder M, Bohnsack O, Nichol G, Humphrey R, Hodi FS. Guidelines for the evaluation of immune therapy activity in solid tumors: immune-related response criteria. Clin Cancer Res. 2009 Dec 1;15(23):7412-20. doi: 10.1158/1078-0432.CCR-09-1624. Epub 2009 Nov 24. PMID 19934295
- [Derived] Arrieta O, Barron F, Ramirez-Tirado LA, Zatarain-Barron ZL, Cardona AF, Diaz-Garcia D, Yamamoto Ramos M, Mota-Vega B, Carmona A, Peralta Alvarez MP, Bautista Y, Aldaco F, Gerson R, Rolfo C, Rosell R. Efficacy and Safety of Pembrolizumab Plus Docetaxel vs Docetaxel Alone in Patients With Previously Treated Advanced Non-Small Cell Lung Cancer: The PROLUNG Phase 2 Randomized Clinical Trial. JAMA Oncol. 2020 Jun 1;6(6):856-864. doi: 10.1001/jamaoncol.2020.0409. PMID 32271354

RESULTS

PARTICIPANT FLOW:
Groups:
- Docetaxel + MK-3475: Docetaxel 75 mg/m2 day 1 every 3 weeks for 6 cycles MK-3475 (200mg, Day 8, every 3 weeks), followed by maintenance therapy with MK-3475 until disease progression or unacceptable toxicity.
- Docetaxel: Docetaxel 75 mg/m2 day 1 every 3 weeks for 6 cycles.
Period: Overall Study
Arm/Group | Docetaxel + MK-3475 | Docetaxel
Started | 40 | 38
Completed | 40 | 38
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Docetaxel + MK-3475 | Docetaxel | Total
Number analyzed (Participants) | 40 | 38 | 78
Age, Continuous [Mean (Standard Deviation); unit: Years] | 50.1 (13.2) | 62.1 (11.6) | 60.01 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 25 | 46
  Male | 19 | 13 | 32
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Mexico | 40 | 38 | 78

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: The objective response rate (ORR) per response evaluation criteria in solit tumors (RECIST v1.1) was defined as the sum of complete response or partial response assessed by RECIST (v1.1) and is presented as the percent of participants with 95% Confidence Intervals (CI). Complete response (CR) was considered if there was a dissapearance of all target lesions, any pathological lymph nodes (whether target or non-target) must have had a reduction in short axis to <10 mm. Partial response (PR) was considered if there was at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. ORR = CR + PR.
Time Frame: from baseline to 2 months of treatment
Measure: Number (95% Confidence Interval); unit: percentage of responders
Arm/Group | Docetaxel + MK-3475 | Docetaxel
Number analyzed (Participants) | 40 | 38
percentage of responders | 42.5 [26.9 to 58.1] | 15.8 [4.0 to 27.6]

ADVERSE EVENTS:
Time Frame: 1 year
Description: All adverse events were recorded during each clinical visit
Groups:
- Docetaxel + MK-3475: Docetaxel 75 mg/m2 every 3 weeks until progression of disease
  MK-3475 (administered on day 8) 200mg every 3 until progression of disease
  MK-3475: The dosing interval of pembrolizumab can be increased in case of toxicity.
  Docetaxel: Use on both arms as standard of care.
Arm/Group | Docetaxel + MK-3475 | Docetaxel
All-Cause Mortality (participants affected / at risk) | 21/40 | 17/38
Serious Adverse Events (participants affected / at risk) | 5/40 | 3/38
Other Adverse Events (participants affected / at risk) | 37/40 | 35/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Docetaxel + MK-3475 (N=40) | Docetaxel (N=38)
Fatigue (General disorders) | 2 (2) | 2 (2)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hyponatremia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hypothiroidism (Endocrine disorders) | 1 (1) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Docetaxel + MK-3475 (N=40) | Docetaxel (N=38)
Fatigue (General disorders) | 26 (26) | 24 (24)
Anemia (Blood and lymphatic system disorders) | 26 (26) | 19 (19)
Nausea (Gastrointestinal disorders) | 21 (21) | 18 (18)
Diarrhea (Gastrointestinal disorders) | 19 (19) | 19 (19)
Neuropathy (Nervous system disorders) | 16 (16) | 18 (18)
Neutropenia (Blood and lymphatic system disorders) | 16 (16) | 15 (15)
Alopecia (Skin and subcutaneous tissue disorders) | 10 (10) | 8 (8)
Vomiting (Gastrointestinal disorders) | 9 (9) | 9 (9)
Hyporexia (Metabolism and nutrition disorders) | 8 (8) | 8 (8)
Lymphopenia (Blood and lymphatic system disorders) | 8 (8) | 0 (0)
Mucositis (General disorders) | 7 (7) | 4 (4)
Constipation (Gastrointestinal disorders) | 6 (6) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 5 (5) | 2 (2)
Hyponatremia (Endocrine disorders) | 4 (4) | 4 (4)
Edema (Skin and subcutaneous tissue disorders) | 4 (4) | 2 (2)
Dysgeusia (Metabolism and nutrition disorders) | 4 (4) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 3 (3)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Hypercalcemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Hyperbilirrubinemia (Hepatobiliary disorders) | 1 (1) | 1 (1)
Hand Foot Syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Lacrimal obstruction (Eye disorders) | 1 (1) | 1 (1)
Paronychia (General disorders) | 1 (1) | 0 (0)
Hypomagnesemia (General disorders) | 0 (0) | 7 (7)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypothiroidism (Endocrine disorders) | 11 (11) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 2 (2)
Hepatitis (Hepatobiliary disorders) | 7 (7) | 4 (4)
Hyperthiroidism (Endocrine disorders) | 3 (3) | 0 (0)
Xerostomy (Immune system disorders) | 2 (2) | 1 (1)
Nephritis (Renal and urinary disorders) | 1 (1) | 1 (1)
Sjogren (Eye disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The data here presented should be interpreted in light of its limitations. Foremost, the study was designed in the absence of recently established information, and therefore, several factors were not available during the patient selection process, including PD-L1 expression for all included patients. Additionally, patients with common oncogenic driver mutations, including EGFR could be enrolled. This generates a heterogeneous population with several already characterized subgroups present.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-21): https://cdn.clinicaltrials.gov/large-docs/98/NCT02574598/Prot_SAP_000.pdf